CLINICAL TRIAL: NCT06805630
Title: Urine-based Methylation Markers in the Diagnosis and Surveillance of Upper Tract Urothelial Carcinoma
Brief Title: Urine Methylation Markers in UTUC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00116347
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-02

CONDITIONS: Upper Tract Urothelial Cancer
Keywords: UTUC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients with primary UTUC (upper tract urothelial carcinoma) (Other): Urine DNA samples will be quantified using Bladder CARE™ at baseline, 3 months, and 6 months.
  Interventions: Diagnostic Test: Bladder CARE™

INTERVENTIONS:
Diagnostic Test: Bladder CARE™ — Urine methylation biomarker test

SUMMARY:
This is a research study to measure DNA markers in the urine of patients with upper tract urothelial cancer (UTUC) before surgery and during follow-up visits. Identifying these DNA markers could improve diagnosis before surgery, help assess risk, and predict early recurrence of the cancer. Urine samples will be de-identified and sent to Pangea Laboratory LLC for analysis. The results of this test will be compared to the traditional tests in upper tract urothelial cancer, such as cells in the urine and tissue biopsy.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years
* Primary UTUC

Exclusion Criteria:

* Patients who do not understand and/or are unwilling to sign a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Methylation level of urothelial-specific biomarker TRNA-Cys | Baseline, 3 months, 6 months
Methylation level of urothelial-specific biomarker SIM2 | Baseline, 3 months, 6 months
Methylation level of urothelial-specific biomarker NKX1-1 | Baseline, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Abern, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No